CLINICAL TRIAL: NCT01233336
Title: Hepatocyte Growth Factor as an Early Marker of Myocardial Injury and Prognostic Factor of Cardiovascular Events in Log-term Follow up in Patients With Acute Coronary Syndrome
Brief Title: Hepatocyte Growth Factor (HGF) Concentration in Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Responsible Party: Sponsor
Other Study IDs: 2.52/VII/10
Record Dates: First submitted 2010-11-02; First posted 2010-11-03 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Acute Coronary Syndrome; Myocardial Infarction
Keywords: ACS,; HGF,; myocardial infarction; markers of myocardial injury; acute coronary syndrome (ACS); prognostic factors in patients with ACS
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma for HGF concentration
Oversight: Data Monitoring Committee: No

SUMMARY:
This is the continuation of previous study (registration number: NCT00844987) which revealed that hepatocyte growth factor (HGF) is a very early, good marker of myocardial injury and prognostic factor for post myocardial infarction (MI) cardiovascular events presence in long-term follow-up. Due to potentially very important implication of the results of previous study it was decided to continue research of HGF in patients with MI. Now, is scheduled to examine 100 consecutive patients with STEMI. HGF assessments will be performed just after admission to hospital, 1h and 24h later and before discharge. Two follow-up visits were planned i.e. at 3 and 6 months after MI. During hospitalization and at 6 month visit the echocardiography examination will be performed. The composite primary endpoint consists of cardiovascular events observed during hospital course and in long term-follow-up.

DETAILED DESCRIPTION:
Hepatocyte growth factor (HGF) was examined in study number NCT00844987 as a potentially useful marker of acute myocardial injury. Results of the study confirmed efficacy of HGF as very early marker of myocardial necrosis and as a prognostic factor for cardiovascular events in long term follow up. Recent study is a continuation of previous study.

The aim is to confirm that maximal values of the HGF in first examination performed in ACS (acute coronary syndrome) patients and to show predictive value of HGF for early and late outcome in patients with ACS.

Materials and method: 100 patients with acute coronary syndrome will be included into the study. HGF will be examined four times i.e. just after admission, 1h and 24h latter and before discharge. In case of 10 patients will be performed 10 assessments during first day of ACS.

The follow up visits will take place 3 and 6 months after ACS. During hospitalization and 6 months later echocardiography examination will be performed and the extension of heart dysfunction will be assessed. Control group will consist of 10-15 health volunteers.

The primary endpoint is a composite endpoint which will include following cardiovascular events observed during hospitalization and during 6-month follow up: death, reinfarction, coronary interventions (PCI and/or CABG) due to new ACS or exacerbation of angina, symptoms of heart failure, rehospitalization due to cardiovascular events and stroke in context of HGF concentration in acute stage of ACS.

As a secondary endpoints will be considered: 1) death, 2) symptoms of heart failure 3)rehospitalization due to cardiac events observed during hospitalization or in 6-month follow-up. All this endpoints will consider in context of HGF values and values of routinely measured markers of myocardial injury.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years,
* chest pain,
* symptoms of ischemia at ECG,
* signed informed consent form

Exclusion Criteria:

* age < 18 years,
* not signed informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with acute coronary syndrome admitted to CCU due to symptoms of ACS.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2010-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
composite end point | 6-month follow -up
  death, reinfarction, coronary interventions (PCI and/or CABG) due to new ACS or exacerbation of angina, symptoms of heart failure, rehospitalisation due to cardiovascular events and stroke in context of HGF concentration in acute stage of ACS

SECONDARY OUTCOMES:
death | 6- month follow-up
  endpoint in context of HGF concentration in early stage of ACS
symptoms of heart failure | 6-month follow-up
  endpoint in context of HGF concentrationin early stage of ACS
rehospitalisation due to cardiovascular reasons | 6- month follow-up
  endpoint in context of HGF concentration in early stage of ACS

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Cardiology , CCU, ul. Alpejska 42, Warsaw, Poland